CLINICAL TRIAL: NCT04747262
Title: Administering a Parent-based Pilot Intervention- SPACE for Reducing Anxiety in Children With ASD
Brief Title: Administering a Parent-based Pilot Intervention for Reducing Anxiety in Children With ASD and Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Analia Shefer, Ph.D, Hebrew University of Jerusalem
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: School of Education /SPACE
Record Dates: First submitted 2021-02-06; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: ASD, Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The program contains 12 weekly 1-hour sessions with the parents. We will examine the impact of the intervention on family accommodation, ASD and anxiety symptomology, as well as parent and child satisfaction from the intervention, using the attached measures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPACE INTERVENTION (Experimental): counseling
  Interventions: Behavioral: SPACE

INTERVENTIONS:
Behavioral: SPACE — SPACE program, an evidence-based protocol that has been proven to be efficent in childhood anxiety disorders and OCD (Lebowitz, 2013; Lebowitz, Omer, Hermes & Scahill, 2014)

SUMMARY:
We are implementing the SPACE program, an evidence-based protocol that has been proven to be efficent in childhood anxiety disorders and OCD (Lebowitz, 2013; Lebowitz, Omer, Hermes & Scahill, 2014), in a new population of children with ASD and anxiety. The intervention aims to reduce family accommodation of the child's anxiety symptoms. The program contains 12 weekly 1-hour sessions with the parents. We will examine the impact of the intervention on family accommodation, ASD and anxiety symptomology, as well as parent and child satisfaction from the intervention, using the attached measures.

DETAILED DESCRIPTION:
Participants are parents of children with ASD and anxiety between the ages of 6-10.

We will recruit 30 families. Recruitment takes place through social media, the Autism Center of Hebrew University, lab contacts and community partnerships. Participants are parents of young children between the ages of 6-10, where the child has a recognized diagnosis of ASD by Ministry of Health, Social Security or Ministry of Education, average (or above) cognition as per parent report and communication as measured by ABAS, and anxiety as measured by SCARED. Parents of children who have other relevant neurological or medical conditions will be excluded. Participants will be asked to provide a copy of the latest diagnosis prior to participation. Measures (attached) will be administered prior to the intervention, at the conclusion and again 2 months later. Participants will complete questionnaires online (Qualtrics). Treatment sessions will be held on ZOOM and certain sessions will be taped for supervision purposes.

The program is designed to reduce child anxiety symptoms, parent stress and family accommodation. Parents are likely to gain important skills and experience an increase in feelings of self-efficacy. The SPACE program is parent-based and is applicable in cases where children are not cooperative, and if proven to be effective in the ASD population, could serve not only as an alternative treatment but also as a primary intervention in the context of ASD..

ELIGIBILITY:
Inclusion Criteria ASD Anxiety Symptoms

Exclusion Criteria:

* Anxiety treatment

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-01-17 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The psychometric properties of the Screen for Child Anxiety Related Disorders (SCARED) are discussed in Birmaher, B., Brent, D. A., Chiappetta, L., Bridge, J., Monga, S., & Baugher, M. (1999). | 15 minutres
  The Screen for Child Anxiety Related Disorders (SCARED) is a 41-item inventory rated on a 3 point Likert-type scale. It comes in two versions; one asks questions to parents about their child and the other asks these same questions to the child directly. The purpose of the instrument is to screen for signs of anxiety disorders in children.
Family Accommodation Scale - Anxiety (FASA) | 15 minutres
  study accommodation across childhood anxiety disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Hebrew university, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rozenblat S, Shimshoni Y, Lebowitz ER, Perez M, Koller J. A Pilot Trial of SPACE (Supportive Parenting for Anxious Childhood Emotions) in Autism. Child Psychiatry Hum Dev. 2025 Feb;56(1):249-263. doi: 10.1007/s10578-023-01555-4. Epub 2023 Jun 23. PMID 37353645